CLINICAL TRIAL: NCT04525482
Title: Application of Early Goal-directed Sedation in Patients With Severe Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-081
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Brain Injuries, Traumatic
Keywords: Brain Injuries; Early Goal-directed Sedation
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention was implemented
- Intervention Group (Experimental): Early goal-directed sedation programs was implemented
  Interventions: Other: Early goal-directed sedation programs

INTERVENTIONS:
Other: Early goal-directed sedation programs — A. Provide sedation at the beginning of the titration of dextrometomidine; b. Optimize sedation when dextrometomidine is used alone and at a maximum dose not sufficient to provide comfort and safety to the patient and to achieve a level of sedation at any time specified by the treating physician. C. Provides immediate recovery and sedation, and can control sudden agitation at any time
  Arms: Intervention Group

SUMMARY:
EGDS management strategy was implemented in ICU patients with severe brain injury, the depth of sedation and GCS score were monitored, and the protective effects of EGDS strategy and standard sedation strategy on the brain of patients with severe brain injury were discussed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe craniocerebral injury
* The GCS score is 6 to 12 points
* Within 12 hours of intubation
* The mechanical ventilation time is greater than 24 hours
* Obtain written consent

Exclusion Criteria:

* Pregnant women
* Acute liver failure
* Dementia or mental illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Richmond Agitation-Sedation Scale | through study completion, an average of 2 year
Mechanical ventilation time | through study completion, an average of 2 year
length of stay in ICU | through study completion, an average of 2 year

SECONDARY OUTCOMES:
complication | through study completion, an average of 2 year

IPD SHARING:
Plan to Share IPD: No